CLINICAL TRIAL: NCT04325542
Title: Prevalence of HBV in Pregnant Women Attending Antenatal Care in Tanzania A Survey on the Prevalence of HBsAg in Pregnant Women in the Region of Mwanza, Tanzania
Brief Title: Prevalence of HBV in Pregnant Women Attending Antenatal Care in Tanzania
Acronym: HBVPMTCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Mission Institute, Germany (Other)
Collaborators: Catholic University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, Dr. Christa Kasang, Research Coordinator, Medical Mission Institute, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HBVPMTCT
Record Dates: First submitted 2019-11-14; First posted 2020-03-27 (Actual); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Hepatitis B
Keywords: Hepatitis B in pregancy; Hepatitis B vertical transmission; Hepatitis B Tanzania; Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Intervention Model Description: Hepatitis B prevalence study of woman attending antenatal care
Oversight: Data Monitoring Committee: No

ARMS (1):
- HBSAG positive with rapid test (Other): Newborns from woman who are positive with HBSAG rapid test got WHO recommended HBV vaccination at birth to avoid HBV transmission
  Interventions: Diagnostic Test: HBSAg (sure screen test)

INTERVENTIONS:
Diagnostic Test: HBSAg (sure screen test) — Diagnostic test for Hepatitis B

SUMMARY:
Chronic Hepatitis B virus (HBV) infection is a neglected disease with devastating consequences, particularly in countries with limited resources for the health sector. Mother-to-child-transmission (MTCT) is responsible for around 50 % of the HBV infections in Tanzania which, in 90 % of the cases, lead to a chronic HBV infection of the child. This infection rate could be reduced with an active immunization directly after birth which is recommended by the World Health Organization (WHO). However, the Tanzanian national immunization programme schedules the first Hepatitis B vaccination for the fourth week after birth which is too late to prevent a perinatal transmission.

The aim of the study is to determine the prevalence of Hepatitis B surface antigen (HBsAg) in pregnant women in rural and urban study sites in the region of Mwanza, Tanzania. The blood from the positive -testing mothers should be further examined for viral load, genotype of the virus and for liver transaminases in order to conceive a better understanding of the progression of the infection. Beside the laboratory parameters, risk factors for the infection should be determined with the use of a questionnaire.

Furthermore we would like to assess the number of children who were already infected, during the intrauterine period or during birth.

DETAILED DESCRIPTION:
Worldwide, more than 2 billion people are infected with hepatitis B virus (HBV). Of these, 240 million are chronic carriers of HBV and are at risk of death from acute fulminant liver disease, liver cirrhosis or hepatocellular carcinoma (HCC). The World Health Organization (WHO) has stated that the prevalence of hepatitis B is highest in sub-Saharan Africa and East Asia and estimates that between 5-10% of the adult population are chronically infected. Currently, several drugs have been approved in industrialized countries for treating chronic HBV infection and these follow established guidelines from professional medical organizations. Antiviral treatment of chronic hepatitis B infection significantly delays the progression of cirrhosis, reduces the incidence of HCC and improves long-term survival. However, in many resource-constrained settings, including Tanzania, the implementation of this treatment has not yet occurred.

The lack of treatment opportunities in resource-constrained settings means that the prevention of HBV infection is crucial. In countries with high HBV prevalence, most HBV transmission occurs during childhood.

In Tanzania, the prevalence of acute or chronic HBV infection (as defined by a positive hepatitis B surface antigen, HBsAg, test) among blood donors or adults in Dar es Salaam, Tanzania was found to be 8.8% and 6%, respectively. People suffering from chronic HBV have a lifelong risk of developing complications like liver cirrhosis, liver failure or hepatocellular carcinoma (HCC). Chronic hepatitis B infection is the main cause for HCC in Tanzania and there is no therapy available. There are no national recommendations or vaccination program against HBV for HCWs in Tanzania. However, in 2002,Tanzania implemented the WHO policy of general HBV vaccination for children as part of the extended program on immunization (known as EPI). According to notified data, a vaccination coverage of 84% among one year-old children was achieved in 2008 with an immunization schedule of 4, 8, 12 weeks after birth . Above 60% of the infections are acquired in the early childhood by transmission from mother to newborn. This early transmission leads to a chronic Hepatitis B infection among 90% of the infected newborn and, therefore, a vaccination at the earliest 4 weeks after birth might be too late to prevent MTCT. As a matter of fact, in Tanzania, we can estimate 1.4 million chronic Hepatitis B infections through mother-to- child transmission in early phase.

There are two interventions that could prevent MTCT:

1. Implementation of Hepatitis B Immunoglobulin (HBIg) to the child directly after birth
2. Active immunization against HBV within 24 hours after birth. The first intervention is very expensive (100€/per child) and is therefore not sustainable for the Tanzanian health system. The second intervention is cheaper and recommended by the WHO.

HBV infection is a neglected disease in low income countries and has been rarely studied in Tanzania. One of the main ways of infection is MTCT and there are several ideas on how to reduce the transmission. Antiviral drugs for infected pregnant women, implementation of HBIg directly after birth or active immunization within 24 hours after birth are the most popular approaches. Unfortunately, none of these is yet implemented in Tanzania due to several reasons. The cost of all the interventions is one argument against their implementation despite the fact that prevention of the infection was proven more cost efficient rather than facing the long-term costs of people suffering from the disease. Another problem is the insufficient knowledge about this topic in the Tanzanian context. More studies with a larger population are necessary to show the importance of an early intervention and the problem resulting from a vaccination happening too late for the cases of MTCT.

Each avoided infection is a benefit for the whole population, as there is a reduced possibility for other children or family members to get infected. To identify the infants at risk a screening program is needed. Therefore, rapid HBsAg tests should be offered for every pregnant woman at public health facilities. With better information, the awareness about the disease improves and the number of fully vaccinated children rises.

In our study we would like to determine the prevalence of HBsAg in pregnant women attending the antenatal clinic in a tertiary hospital, a regional hospital or a district hospital in Tanzania. The study population should be identified with an HBsAg rapid test at the department of gynaecology. Blood will be taken from the mothers with positive HBsAg rapid test and from the cord blood of their children. Furthermore, we want to assess the risk factors that might lead to an increased risk of hepatitis B infection. Therefore, our research assistants will inquire among the participants about several risk factors. To give some benefit to the patient, we will vaccinate the child of HBsAg positive mothers within 24 hours after birth with an active immunization which is proven to reduce the possibility of MCTC.

The laboratory examination of the blood will give us more details about the serology, genotype and viral load of the HBV infection. This might show us the relation between the risk factors and possible intrauterine HBV transmission.

In Tanzania, there is not enough data on prevalence, risk factors, viral load and genotypes of HBV. This study will give additional data on intrauterine infection of the children.

The general objective of the study is to determine the prevalence of Hepatitis B surface antigen (HBsAg) in women attending antenatal clinic in four different study sites in the region of Mwanza, Tanzania.

Specific objectives are:

1. To determine the viral load and genotype of HBV infection in pregnant woman.
2. To determine the risk factors associated with HBV infections in pregnant women.
3. To determine the prevalence of intrauterine infection by positive HBV PCR of cord blood of the children of HBsAg positive mothers attending BMC, Seka Toure or Sengerema hospital for delivery.
4. To determine the influence of HBV genotypes, viral load and HBeAg status of the mother attending BMC for delivery on the probability of the transmission to the child.

Methodology

The study will be conducted in three different study sites:

In the Department of Obstetrics and Gynaecology of the Bugando Medical Center (BMC) in Mwanza, Tanzania. The department has every year 6000 deliveries, for the second part of the study we choose only the HBsAg positive women diagnosed with a rapid test.

The second sites will be the Mwanza regional hospital Seka Toure and the third will be the district hospital in Sengerema. About 500 woman will be tested in BMC and 250 women will be tested on each other study site, Altogether 1000 patients

Collaborating Institutions are the BMC, and the Catholic University of Health and Allied Sciences (CUHAS) in Mwanza, Tanzania, the division of Medical Virology, Faculty of Medicine & Health Sciences, Stellenbosch University and NHLS Tygerberg, Cape Town, South Africa, the Medical Mission Institute and the University of Würzburg/Institute of Virology and Immunobiology, Würzburg, Germany.

Study design:

The study is a cross-sectional study.

Study patient groups:

Pregnant women aged 18 years and above attending the antenatal clinics at Bugando Medical Center, regional hospital Seka Toure and district hospital in Sengerema.

Sample size For a cross-sectional study sample size was calculated with an expected prevalence of 3,5 % based on previous studies (17).

Level of significance = 5%, Power = 80%, Type of test = cross-sectional Formula of calculating sample size is (38) n = [Z1-α/2²p(1-p)]/d²

We are planning a study of 1000 woman. If the true prevalence is 3.5 % we will need to study at least 51.9 patients to be able to reject the null hypothesis that the exposure rates for case and controls are equal with probability (power) 0.8.

Sample collection and duration To diagnose the hepatitis B positive mothers, a finger prick test will be conducted with pregnant women to assess whether there is HBsAg or not. If the test is positive, 12 ml of EDTA-blood will be taken (3 times 4 ml)), centrifuged and plasma will be stored at -20°C for further analysis.

For the second part of the study, cord blood of children born at the BMC 1.5 ml will be collected after birth and stored at -20°C for further analysis. After 24 months, another blood sample will be taken and stored at -20°C for further analysis. The blood from all HBsAg positive mothers will be analysed including serology for Hepatitis B (HBsAg, HBeAg), HBV-DNA PCR and liver transaminases for the women from the primary health care clinics. The blood from the children will be analysed with HBV-DNA PCR. Taking cord blood and proceeding it immediately after birth will be logistical only possible in BMC so that these analyses will be done in the children born at the BMC and not of the other study sites.

The questionnaire and blood samples will be labelled with the study number only.

Data Collection A questionnaire will used to collect information concerning the risk factors information, including HIV status, age, residence, marital status, level of education, occupation, parity and gravity, history of life-time sexual partners, age at first sexual contact, history of risk factors (blood transfusion, operation, drug use, iv injection), HBV vaccination, history of STIs, condom use, genital circumcision, sharing toothbrush or razors and history of jaundice in the family or for themselves (Case report form). The patients' data will be collected at the time of the enrolment. CRF forms will be supplied. These forms must be printed legibly. A copy will remain at the investigator's files. CRF and all original data should be readily available for review during scheduled monitoring visits. For patient identification, all patients included in the study will have their hospital record number, their date of birth and a patient allocation number entered chronologically into the study file. Copies of all pertinent information will be retained by the investigator for a period of at least 10 years after study completion.

Laboratory Analyses Analysis of the blood On the day of enrolment, a point-of-care Hepatitis B surface antibody tests will be performed. The test (Nal Diagnostics) is CE certified. According to data of the manufacturer, sensitivity, specificity and accuracy of the test are > 99% with a cut off value of m10 IU anti-HBs.

Plasma samples will be frozen at -20°C and shipped for further analysis after enrolment is completed. In the Division of Medical Virology, University of Stellenbosch, the following tests will be carried out for all samples using ELISA-techniques for serological testing and PCR for viral load measurements:

* Hepatitis B - surface antigen (HBsAg)
* Hepatitis B - surface antibody (anti-HBs)
* Hepatitis B - core antibodies (anti-HBc)

This test panel will allow differentiation between naturally-acquired infection, antibodies due to vaccination and chronic hepatitis B.

Cases of chronic hepatitis B will undergo further testing for:

* Hepatitis B e- antigen (HBeAg)
* Hepatitis B e- antibodies (anti-HBe)

For HBV DNA PCR, the DNA will be isolated from the plasma by the column extraction method and PCR amplification will be carried out. A positive PCR reaction will be sequenced with the ABI-Prism-310-Genetic-Analyzer-System. Sequences will be submitted to GenBank. With these methods.

* Hepatitis B viral load
* Hepatitis B genotyping

will be determined. To detect the amount of liver transaminases in the plasma, it will be analysed with spectrophotometric measurements for

* Aspartate aminotransferase (AST/GOT)
* Alanine aminotransferase (ALT/GPT) Statistical Analysis The entries of the Questionnaire will be transferred to an EXCEL Sheet by double entry. The second entry will be completed timely independently from the first entry and will be compared with the first entry. P < 0.05 will be considered as statistically different. The 95% confidence intervals (CI) will be calculated using SPSS and GraphPad Prism Software.

Ethical considerations Ethical committee/institutional review board The final approved protocol including the informed consent form will be submitted for Ethical Clearance to the joint Bugando Medical Centre/Catholic University of Health and Allied Sciences (BMC/CUHAS) Ethics and Review Committee. The investigator will agree to make required progress reports to the Ethics and Review committee, as well as report any serious adverse events, life-threatening problems or deaths. The Ethics Committee/ must be informed by the investigator of the termination of the study. Permission will be sought from the relevant authorities of the study sites clinics.

Patient informed consent Prior to inclusion into the study, the patient will be informed of the nature of the study and will be given pertinent information as to the intended purpose, possible benefits, and possible adverse experiences. The procedure and possible hazards to which the patient is exposed will be explained. An informed consent statement will then be read and signed by the patient, a witness, and the investigator.

Possible benefits for the patients Directly after birth, vaccination is one of the most effective methods to reduce the Hepatitis B transmission from the infected mother to her child. Our study will give all the pregnant women the opportunity to do a rapid test free of any costs. If it is positive, the mother can protect the new-born child from HBV infection via active immunization (in case she will give birth at the study site. and the devastating consequences with a free of cost follow-up screening at the BMC.

Even though the women themselves cannot get any treatment for their disease, the diagnosis may increase their awareness of this infection and possibly contribute to the reduction of transmission.

The child born at the study site gets the benefit of an extra protection with the vaccination directly after birth.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above.
* Signed consent form

Exclusion Criteria:

* Psychiatric disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2018-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Kalluvya, Prof, Principal Investigator — Bugando Medical Center
Locations (1):
- Bugando Medical Center, Mwanza, Tanzania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HBSAG Positive With Rapid Test
Started | 743 (one participant withdraw consent during the study)
Completed | 742
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | HBSAG Positive With Rapid Test
Number analyzed (Participants) | 742
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 742
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [22 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 742
  Male | 0
Region of Enrollment [Number; unit: participants]
  Tanzania | 742

OUTCOME MEASURES:

1. Primary Outcome: HBsAG Prevalence
Description: Number of women attending antenatal clinic at the Bugando Medical Center in Mwanza, Tanzania with Hepatitis B surface antigen (HBsAg) rapid test positive result.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- HBSAG Positive With Rapid Test: Number of women attending antenatal clinic at the Bugando Medical Center in Mwanza, Tanzania with Hepatitis B surface antigen (HBsAg) rapid test positive result.
  HBSAg (sure screen test): Diagnostic test for Hepatitis B
Arm/Group | HBSAG Positive With Rapid Test
Number analyzed (Participants) | 743
Participants | 22

ADVERSE EVENTS:
Time Frame: Adverse events were only collected during the process. It was only blood taken and a finger prick. No intervention was given in this study. So only on Day 1
Description: Adverse events were only collected during the process. It was only blood taken and a finger prick. No intervention was given in this study. So only on Day 1
Arm/Group | HBSAG Positive With Rapid Test
All-Cause Mortality (participants affected / at risk) | 0/742
Serious Adverse Events (participants affected / at risk) | 0/742
Other Adverse Events (participants affected / at risk) | 0/742

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No